CLINICAL TRIAL: NCT03042273
Title: A Randomised, Double-blind, Placebo Controlled Study to Investigate the Efficacy and Safety of High Strength Cranberry (Pacran®) in Women With Recurrent Urinary Tract Infections (Cystitis)
Brief Title: High Strength Cranberry Supplementation for Prevention of Recurrent Urinary Tract Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swisse Wellness Pty Ltd (Industry)
Collaborators: Commonwealth Scientific and Industrial Research Organisation, Australia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PAC-001
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2019-06

CONDITIONS: Urinary Tract Infection
Keywords: recurrent
MeSH Terms: conditions — Urinary Tract Infections; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Strength Cranberry (Experimental): 1 capsule of High Strength Cranberry (25,000mg Vaccinium macrocarpon) orally daily for 6 months
  Interventions: Dietary Supplement: High Strength Cranberry
- Placebo (Placebo Comparator): 1 capsule of Matching Placebo orally daily for 6 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: High Strength Cranberry — Softgel capsule
  Other Names: 25,000mg Vaccinium macrocarpon
  Arms: High Strength Cranberry
Dietary Supplement: Placebo — Soy oil to match High Strength Cranberry Softgel Capsule
  Other Names: Placebo (for High Strength Cranberry)
  Arms: Placebo

SUMMARY:
This clinical trial is a Phase 2, multicenter, placebo-controlled, double-blind, parallel-arm study to evaluate the efficacy and safety of High Strength Cranberry (500mg Pacran®) in preventing UTI (cystitis) in women with a history of recurrent UTI (rUTI).

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18-65 years, inclusive
2. A history of recurrent urinary tract infection defined as ≥3 UTIs in the last year OR at least 2 UTIs occurring in the last 6 months. Each infection requires confirmation by a health professional
3. Willing to answer questionnaires and comply with the study requirements
4. Ability to swallow capsules
5. Provided Written Informed Consent
6. BMI >17.5kg m2 and <35kg m2

Exclusion Criteria:

1. Microbial growth on urine culture of ≥107 cfu/L (104cfu/mL) within 7 days of Day 1
2. A history of >5 UTIs in the last 6 months (confirmed by self-report or health professional)
3. Use of antibiotics or antibiotics for prophylaxis within 28 days of Day 1
4. Use of any antibacterial products, that in the opinion of the Medical Investigator may interfere with the study outcomes, within 28 days of Day 1
5. Regular use of Vaccinium containing products (e.g. all forms of blueberries, cranberries, bilberry, lingonberry , etc i.e fruit, dried fruit, pills, juices or supplements) within 28 days of Day 1 at the discretion of the Medical Investigator
6. Presence of an intermittent or indwelling urinary catheter
7. Anatomical abnormalities of the urinary tract
8. History of or known clinically significant renal or urological disease(self-reported)
9. Positive urine dipstick pregnancy test at screening onDay 1, currently pregnant and/or breastfeeding
10. Women of Childbearing potential not willing to use adequate and effective methods of contraception throughout the study
11. Women of child bearing potential that have not been using effective methods of contraception for 14 days prior to Day 1
12. History of or known clinically significant cardiac disease
13. History of or known clinically significant liver disease
14. History of or known clinically significant gastrointestinal disease
15. History of or known metabolic disorder or diabetes
16. History or presence of alcohol or illicit drug abuse,any surgical history, clinical condition or organ dysfunction that in the opinion of the Medical Investigator may affect the participant's ability to participate in the study or the study results
17. Currently hospitalised or any planned hospitalisations within 1 month following the last dose of study product
18. Immunocompromised participants or participants receiving immunosuppressive medication
19. History of an adverse reaction or known hypersensitivity or suspected allergy to the investigational product ingredients
20. Currently taking warfarin or has received Warfarin within 28 days of Day 1
21. Received an investigational drug within 28 days of Day 1

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with a history of recurrent UTIs
Enrollment: 150 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of UTI | 6 months
  cultured confirmed UTIs at a level of >108cfu/L (105cfu/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Welma Stonehouse, PhD, Principal Investigator — Commonwealth Scientific and Industrial Research Organisation, Australia
Locations (5):
- Australia (5):
  - Holdsworth House Medical Centre, Sydney, New South Wales
  - Holdsworth House Medical Centre, Brisbane, Queensland
  - Griffith University Clinical Trial Unit (Griffith Health), Gold Coast, Queensland
  - CSIRO Nutrition and Health Research Clinic, Adelaide, South Australia
  - Monash Alfred Psychiatry Research Centre (MAPrc), Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stonehouse W, Benassi-Evans B, Bednarz J, Vincent AD. Whole cranberry fruit powder supplement reduces the incidence of culture-confirmed urinary tract infections in females with a history of recurrent urinary tract infection: A 6-month multicenter, randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2025 Apr;121(4):932-941. doi: 10.1016/j.ajcnut.2025.01.022. Epub 2025 Jan 23. PMID 39863114